CLINICAL TRIAL: NCT02005705
Title: Randomized Trial of Outpatient vs. Inpatient Management of Low-risk Patients With Upper Gastrointestinal Bleeding.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate recruitment
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Loren Laine, Professor of Medicine, Yale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIC 1307012373
Record Dates: First submitted 2013-12-03; First posted 2013-12-09 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Upper Gastrointestinal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Outpatient (Active Comparator)
  Interventions: Other: Outpatient Management of Low-risk Patients
- Inpatient (Active Comparator)
  Interventions: Other: Inpatient Management of Low-risk Patients

INTERVENTIONS:
Other: Outpatient Management of Low-risk Patients — * Labs will be obtained within 2-3 days of discharge from ED
  * Clinic visit will be scheduled within 3 days of discharge from ED
  * EGD will be scheduled within 7 days of discharge from ED
  * Phone follow-up at day 7 and 30
  Arms: Outpatient
Other: Inpatient Management of Low-risk Patients — * Labs will be obtained on day of discharge or day 2-3
  * EGD will be performed in the hospital
  * Phone follow-up at day 7 and 30
  Arms: Inpatient

SUMMARY:
Patients presenting to the emergency room with upper gastrointestinal bleeding and a Glasgow Blatchford score of zero will be randomly assigned to further care in the inpatient vs. outpatient setting. The hypothesis of this study is that patients who are managed as outpatients will require interventions at a rate not higher than those managed as inpatients and will have lower direct healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

1. Blood Urea Nitrogen < 18.2 mg/dl
2. Hemoglobin ≥ 13.0 g/dl for men and ≥ 12.0 g/dl for women
3. Systolic blood pressure ≥ 110 mm Hg
4. Heart rate < 100 beats/min

Exclusion Criteria:

1. Inability to obtain informed consent
2. Pregnancy
3. History of liver disease
4. History of heart failure
5. Syncope that is temporally related to ongoing bleeding
6. Melena
7. Contraindication to proton pump inhibitor use
8. Other conditions that necessitate inpatient evaluation.
9. Inpatients with new onset of GI bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The number of patients requiring intervention for UGIB (endoscopic therapy, blood transfusion, surgery, interventional radiology) | Within 7 days of the index presentation to the emergency room

CONTACTS AND LOCATIONS:
Overall Officials: Loren Laine, MD, Principal Investigator — Yale University, Section of Digestive Disease
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States